CLINICAL TRIAL: NCT06867640
Title: Effects of Forgiveness-Based Group Psychoeducation Applied to Cancer Survivors on Fear of Cancer Recurrence, Forgiveness and Psychiatric Symptoms: A Randomized Controlled Trial
Brief Title: Effects of Forgiveness-Based Group Psychoeducation Applied to Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hilal Merve Belen (Other Government)
Collaborators: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor-Investigator, Hilal Merve Belen, Principal Investigator, Lokman Hekim University
Organization: Lokman Hekim University (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: LokmanHekimU-HMB-1
Record Dates: First submitted 2025-02-23; First posted 2025-03-10 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-02

CONDITIONS: Cancer Survivors
Keywords: Cancer Survivors; Forgiveness; Psychoeducation; Fear of Cancer Recurrence; Quality of Life; Psychiatric Symptoms

STUDY DESIGN:
Intervention Model Description: Forgiveness-Based Group Psychoeducation
Who Masked: Outcomes Assessor
Masking Description: The process of assigning participants to groups will be carried out by a statistician outside the study using the simple randomization method and will be hidden from the researcher until the application begins. Since the assignment to groups will be made after informed consent is obtained, the participants will be blinded (single blind). In addition, the statistician will also be blinded in order to reduce statistical analysis and reporting bias. Without specifying which group (intervention and control group) the data belong to, they will be coded and transferred to the database (group A, group B), and the data will be analyzed and reported.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Forgiveness-Based Group Psychoeducation (Experimental): Forgiveness-based group psychoeducation to be conducted with the experimental group is planned as 6 sessions. The sessions are planned to be conducted in 3 groups of 8-10 people. The duration of a session is planned to be approximately 90 minutes. Group psychoeducation with the experimental group will be conducted face-to-face every week. The appropriate day for the sessions will be decided with the members of each group. The same group sessions will be conducted on the same day and time every week.
  Interventions: Other: Forgiveness-Based Group Psychoeducation
- No Intervention (No Intervention): After the follow-up tests were completed, it was planned to implement the 6-session forgiveness-based group psychoeducation applied to the intervention group in the same way upon the request of the control group.

INTERVENTIONS:
Other: Forgiveness-Based Group Psychoeducation — The effect of forgiveness-based group psychoeducation applied to cancer survivors on fear of cancer recurrence, forgiveness and psychiatric conditions.
  Arms: Forgiveness-Based Group Psychoeducation

SUMMARY:
This study aims to examine the effects of forgiveness-based group psychoeducation applied to cancer survivors on fear of cancer recurrence, forgiveness and psychiatric symptoms.

DETAILED DESCRIPTION:
This study was designed as a randomized controlled experimental study with a pre-test-post-test and follow-up design to examine the effects of forgiveness-based group psychoeducation on fear of cancer recurrence, forgiveness and psychiatric symptoms of cancer survivors.

The aim is to evaluate the effects of a forgiveness-based psychoeducation program on cancer survivors. After the "Informed Voluntary Consent Form" is obtained from individuals who agree to participate in the study, the Introductory Information Form, Heartland Forgiveness Scale, Fear of Relapse Inventory and Brief Symptom Inventory will be applied. Pre-tests will be applied to the sample determined by an independent statistician. Then, participants will be divided into intervention and control groups by simple randomization method. Face-to-face forgiveness-based psychoeducation will be applied to the intervention group in 90-minute sessions once/twice a week, totaling 6 sessions. In the last session of psychoeducation, a post-test ("Introductory Information Form", "Heartland Forgiveness Scale", "Fear of Relapse Inventory" and "Brief Symptom Inventory") will be administered to both the intervention and control groups. The first follow-up test of the study will be administered to both the intervention and control groups 1 month after the post-test, and the second follow-up test of the study will be administered 3 months after the post-test. After the completion of the study and the measurements, it is planned to provide forgiveness-based psychoeducation to the participants in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Written and verbal consent to participate in the study
* Understanding and speaking Turkish
* Being over 18 years old
* Not having any visual, hearing or mental disabilities
* Having been diagnosed with cancer, treated with curative intent and having completed major treatments (surgery, radiotherapy, chemotherapy) within the last 5 years

Exclusion Criteria:

* Not volunteering to participate in research
* Having a visual, hearing or mental disability
* Agreeing to participate in another psychoeducational program conducted simultaneously with the research
* Inability to communicate in Turkish
* Having previously received training in forgiveness and/or coping with fear of relapse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2025-04-02 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Heartland Forgiveness Scale | Baseline, 6 th week, 1st month follow-up, 3rd month follow-up) (Pre-test-post-test follow-up experimental design)
  The scale, which evaluates the level of forgiveness and consists of 18 items, consists of three sub-dimensions: "forgiveness of self", "forgiveness of others" and "forgiveness of the situation". The items of the Likert-type scale are evaluated according to a 7-point evaluation scale and the evaluation is answered as "does not reflect me at all" (1 point), "does not reflect me very much" (3 points), "reflects me a little" (5 points) and "reflects me completely" (7 points). Items 2, 4, 6, 7, 9, 11, 13, 15 and 17 in the scale items are scored reversely. The scale is evaluated according to total and sub-scale scores and there is no cut-off score. High scores obtained from each of the sub-dimensions of the scale indicate a high or low level of forgiveness in the relevant sub-dimension. The total forgiveness score is formed by summing the scores of the sub-dimensions of the scale.

SECONDARY OUTCOMES:
Brief Symptom Inventory | Baseline, 6th week, 1st month follow-up, 3rd month follow-up) (Pre-test-post-test follow-up experimental design)
  It is a Likert-type scale and the items are scored by rating them between 0 and 4, with the statements "not at all" and "a lot". People who will fill out the scale are asked to read each item separately and indicate how much each of these symptoms has bothered them in the last week, including that day. When the total for each subscale is divided by the number of items in that subscale, a score for that dimension is obtained. Brief Symptom Inventory subscale dimensions and items; anxiety; items 12, 13, 28, 31, 32, 36, 38, 42, 43, 45, 46, 47, 49; depression; items 9, 14, 16, 17, 18, 19, 20, 25, 27, 35, 37, 39; negative self; Items 15, 21, 22, 24, 26, 34, 44, 48, 50, 51, 52, 53; somatization; items 2, 5, 7, 8, 11, 23, 29, 30, 33; hostality; items 1, 3, 4, 6, 10, 40, 41.
Fear of Cancer Recurrence Inventory | Baseline, 6th week, 1st month follow-up, 3rd month follow-up) (Pre-test-post-test follow-up experimental design)
  The scale, which has a five-point Likert structure, consists of 42 items and 7 sub-dimensions. These sub-dimensions are; triggers (items 1-8 and 9-17), psychological distress (items 18-21), functional disorders (items 22-27), insight (items 28-30), self-relaxation methods (items 31-33), coping methods (items 34-42). The scale, which does not have any cut-off point, is scored as 0-4 points. It is obtained by adding the questions in each sub-dimension straight, except for question 43. The total scores that can be obtained from the scale are between 0-168, and as the score increases, it is judged that the fear of relapse increases.

OTHER OUTCOMES:
Introductory Information Form | Baseline, 1st month follow-up, 3rd month follow-up (Pre-test-post-test follow-up experimental design)
  It was created by the researchers in line with the literature information in order to determine the participants' sociodemographic (age, gender, marital status, education level, etc.) and diagnosis-treatment process-related characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Sarıkoç, Associate Professor, Study Director — Saglik Bilimleri Universitesi
Locations (1):
- Gülhane Health Sciences Institute, Ankara, Keçiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No